CLINICAL TRIAL: NCT00030875
Title: A Phase II Study Of PS-341 (NSC 681239) In Patients With Untreated Or Relapsed Mantle Cell Lymphoma
Brief Title: Bortezomib in Treating Patients With Mantle Cell Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NCIC Clinical Trials Group (Network)
Responsible Party: Sponsor
Organization: Canadian Cancer Trials Group (Network)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I150; CAN-NCIC-IND150 (Other: PDQ); CDR0000069207 (Other: PDQ)
Record Dates: First submitted 2002-02-14; First posted 2003-01-27 (Estimated); Last update posted 2023-08-04 (Actual); Status verified 2020-04

CONDITIONS: Lymphoma
Keywords: stage I mantle cell lymphoma; contiguous stage II mantle cell lymphoma; noncontiguous stage II mantle cell lymphoma; stage III mantle cell lymphoma; stage IV mantle cell lymphoma; recurrent mantle cell lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Mantle-Cell | interventions — Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

INTERVENTIONS:
Drug: bortezomib

SUMMARY:
RATIONALE: Bortezomib may stop the growth of cancer cells by blocking the enzymes necessary for cancer cell growth.

PURPOSE: Phase II trial to study the effectiveness of bortezomib in treating patients who have previously untreated or relapsed mantle cell lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the efficacy of bortezomib, in terms of response rate, in patients with previously untreated or relapsed mantle cell lymphoma.
* Determine the toxicity of this drug in these patients.
* Correlate suppression of 20S proteasome levels with toxicity of and response to this drug in these patients.
* Determine the time to progression and response duration in patients treated with this drug.

OUTLINE: This is a nonrandomized, multicenter study.

Patients receive bortezomib IV over 3-5 seconds on days 1, 4, 8, and 11. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity. Patients with complete response (CR) receive 2 courses beyond documentation of CR. Patients with stable disease receive a maximum of 4 courses. Patients with partial response (PR) continue therapy until disease progression or for 2 courses beyond documentation of stable PR.

Patients are followed at 4 weeks and then every 3 months until disease progression.

PROJECTED ACCRUAL: A total of 14-30 patients will be accrued for this study within 18-24 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed relapsed or untreated mantle cell lymphoma

  * No refractory disease defined as progression while on chemotherapy or within 1 month after completion of chemotherapy
* At least 1 bidimensionally measurable disease site*

  * Lymph nodes at least 1.5 cm by 1.5 cm by spiral CT scan OR
  * Non-nodal lesions (e.g., skin lesion or nodules) at least 1 cm by 1 cm by MRI, CT scan, or physical exam NOTE: *Bone lesions are not considered bidimensionally measurable disease
* No pre-existing ascites or pleural effusion
* No known CNS involvement by lymphoma

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2

Life expectancy:

* At least 12 weeks

Hematopoietic:

* Absolute granulocyte count at least 1,500/mm^3
* Platelet count at least 75,000/mm^3

Hepatic:

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* AST or ALT no greater than 2.5 times ULN

Renal:

* Creatinine no greater than 1.5 times ULN

Cardiovascular

* LVEF at least 45% by echocardiogram or MUGA

Pulmonary

* No pre-existing shortness of breath greater than grade 1

Other:

* No uncontrolled bacterial, fungal, or viral infections
* No pre-existing edema greater than grade 1
* No pre-existing neuropathy greater than grade 1
* No other malignancy within the past 5 years except adequately treated nonmelanoma skin cancer or carcinoma in situ of the cervix
* No other serious illness or medical condition that would preclude study compliance
* No geographical conditions that would preclude study compliance
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* See Chemotherapy
* Prior rituximab allowed
* No prior radioactive monoclonal antibody therapy

Chemotherapy:

* See Disease Characteristics
* No prior high-dose chemotherapy with stem cell transplantation
* No more than 2 prior systemic chemotherapy regimens

  * Same chemotherapy combination given for first-line and second-line therapy is considered 2 regimens
* No prior flavopiridol
* At least 6 weeks since prior chemotherapy
* No concurrent cytotoxic chemotherapy

Endocrine therapy:

* No concurrent corticosteroids

Radiotherapy:

* No prior radiotherapy to 25% or more of functioning bone marrow
* At least 4 weeks since prior radiotherapy (except low-dose nonmyelosuppressive radiotherapy) and recovered
* No concurrent radiotherapy to the sole site of measurable disease

Surgery:

* At least 2 weeks since prior major surgery

Other:

* No prior investigational therapy
* No other concurrent anticancer therapy
* No other concurrent investigational anticancer therapy

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2002-11-19 (Actual); Primary Completion 2005-07-21 (Actual); Study Completion 2009-12-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew R. Belch, MD, Study Chair — Cross Cancer Institute at University of Alberta
Locations (10):
- Canada (10):
  - Cross Cancer Institute, Edmonton, Alberta
  - British Columbia Cancer Agency, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Margaret and Charles Juravinski Cancer Centre, Hamilton, Ontario
  - Kingston Regional Cancer Centre, Kingston, Ontario
  - Cancer Care Ontario-London Regional Cancer Centre, London, Ontario
  - Toronto Sunnybrook Regional Cancer Centre, Toronto, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - Maisonneuve-Rosemont Hospital, Montreal, Quebec
  - McGill University, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Belch A, Kouroukis CT, Crump M, Sehn L, Gascoyne RD, Klasa R, Powers J, Wright J, Eisenhauer EA. A phase II study of bortezomib in mantle cell lymphoma: the National Cancer Institute of Canada Clinical Trials Group trial IND.150. Ann Oncol. 2007 Jan;18(1):116-121. doi: 10.1093/annonc/mdl316. Epub 2006 Sep 13. PMID 16971665
- [Result] Belch A, Kouroukis CT, Crump M: Phase II trial of bortezomib in mantle cell lymphoma. [Abstract] Blood 104(11): A-608, 2004.
- [Result] Assouline S, Belch A, Sehn L, et al.: A phase II study of bortezomib in patients with mantle cell lymphoma. [Abstract] Blood 102 (11 Pt 1): A-3358, 2003.